CLINICAL TRIAL: NCT06443931
Title: Cryoablation of Intercostal Nerves for Pain Management in Early Postoperative Period in Patients With Minimally Invasive Mitral Valve Surgery: a Pilot Prospective Randomized Study
Brief Title: Cryoablation of Intercostal Nerves for Pain Management in Early Postoperative Period in Patients With Minimally Invasive Mitral Valve Surgery
Acronym: BLOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-4
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation; Pain, Postoperative
Keywords: cryoablation; pain; minimally invasive mitral valve surgery
MeSH Terms: conditions — Mitral Valve Insufficiency; Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Patients undergoing minimally invasive mitral valve surgery while on cardiopulmonary bypass will be randomized into two groups:
  1. Patients receiving cryoablation of intercostal nerves (CryoINB) as a method of pain relief.
  2. Patients who will undergo a standard pain management protocol.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation of intercostal nerves group (Experimental): Patients in the CryoINB group will undergo cryoablation of the intercostal nerves, at the end of surgery before weaning from CPB, using the "ArtiCue" device for 120 seconds at a temperature of -50°C to -70°C, in the intercostal spaces where the surgical approach is located, one intercostal space above and one below it.
  Interventions: Procedure: cryoablation of intercostal nerves
- Standard pain management protocol group (No Intervention): Patients in the group with the standard anesthesia protocol will receive an intercostal block in the area of surgical access - a single injection of 0.75% ropivacaine solution 20 ml.

INTERVENTIONS:
Procedure: cryoablation of intercostal nerves — Patients in the CryoINB group will undergo cryoablation of the intercostal nerves, at the end of surgery before weaning from CPB, using the "ArtiCue" device for 120 seconds at a temperature of -50°C to -70°C, in the intercostal spaces where the surgical approach is located, one intercostal space above and one below it. Cold leads to axonotmesis, in which the axon and myelin sheath are damaged, preventing the pain signal from traveling along the sensory nerve. However, the structural elements of the nerve are preserved, which promotes complete regeneration at a rate of 1-2 mm per day, thereby restoring normal function within several months.
  Arms: Cryoablation of intercostal nerves group

SUMMARY:
A single-center, pilot, prospective, randomized clinical trial with a 1:1 allocation ratio. The aim of our trial is to determine whether cryoablation of intercostal nerves provides a clinically significant analgesic effect, which is reflected in a decrease in opioid analgesics consumption and in a decrease in pain according to VAS in patients undergoing minimally invasive mitral valve surgery. To obtain preliminary data for planning a subsequent larger prospective randomized trial.

DETAILED DESCRIPTION:
Cardiovascular diseases are one of the main causes of death worldwide. According to pathological studies, heart defects occur in 4-7% of cases, and the most common defect among the defects is damage to the mitral valve. Significant advances in surgical practice, instrumentation, tissue manipulation, and perfusion technology have made it possible to perform mitral valve surgery using mini-approaches. Minimally invasive mitral valve surgery has become the standard of care in some specialized cardiac centers around the world due to its excellent results, even despite longer cardiopulmonary bypass times and aortic occlusion. In 2008 a meta-analysis has been published in which the authors come to the conclusion that a minimally invasive approach for correcting mitral valve pathology actually has significant advantages: early activation of patients, shorter duration of stay in the recovery room, shorter wound healing times, advantages in case of repeated interventions, less the number of bleedings and purulent-septic complications compared to classical sternotomy. But despite all the advantages of this approach, severe pain after minimally invasive cardiac surgery continues to remain a serious problem. Acute pain occurs after dissection of the chest, pleura and pericardium, compression of the intercostal nerve with a retractor, as well as dissection of the intercostal and pectoral muscles during surgical access. It limits breathing and cough in the postoperative period, which can subsequently lead to hypoxemia, sputum stagnation, atelectasis, pneumonia, myocardial ischemia, slow recovery, and also an increase in the length of hospitalization. Therefore, additional emphasis and attention is paid to protocols for early functional restoration and pain reduction for this group of patients. There are protocols for "accelerated recovery after surgery" (ERAS - Enhanced Recovery After Surgery), their use makes it possible to achieve shorter stays in the intensive care unit, reduce hospitalization, improve treatment outcomes and reduce financial costs. One of the components of ERAS is the use of additional pain management modalities. However, in cardiac surgery, traditional methods of regional anesthesia, such as thoracic epidural anesthesia or paravertebral block, are not usually used due to intraoperative heparinization and the associated higher risk of spinal or epidural hematoma. Finding an optimal and effective pain management strategy for this category of patients remains an unsolved problem today.

Intercostal nerve cryoablation is considered a relatively new treatment for postoperative pain in patients undergoing minimally invasive mitral valve surgery. One of the first studies of cryoneurolysis was conducted back in 1974 in thoracic surgery. In 76 patients, the use of intercostal cryoablation resulted in a significant reduction in postoperative opioid analgesic consumption. These results were subsequently confirmed in several other studies and the data were retrospective. In 2000, a prospective randomized controlled trial was published involving 30 patients who underwent minimally invasive mitral valve surgery or minimally invasive coronary artery bypass grafting and underwent intercostal cryoablation. According to the results, a decrease in postoperative pain syndrome was observed, and less painkillers were required.

In the study in patients undergoing surgical stabilization of the ribs, cryoablation of the intercostal nerves resulted in a 25% reduction in opioid analgesics consumption compared with patients who received an extrapleural catheter, and pain scores were reduced by 22% in the cryoablation group. Similar results (cryoablation made it possible to significantly reduce morphine consumption compared to the control group and reduce pain)were also described inrecent retrospective studies through 2023 in other patient groups: patients who have undergone pulmonary resectionusing single-port thoracic video-assisted access, where cryoablation was used as a method of postoperative pain relief and patients undergoing lung transplantation.

In the other study for 2021 the use of this method in patients with lateral thoracotomy showed significant improvement in spirography parameters (FEV1, FVC) after 48 hours, as well as 30 and 60 days after surgery. Studying the influence of pain was not the main objective of this work; pain was assessed using VAS and did not show a difference. However, improvement in breathing parameters in the early postoperative period may indirectly be associated with a lower level of pain and a more comfortable state of the patient; the consumption of opioid analgesics was not properly assessed in this study.

In 2021 published a systematic review of 23 studies on the effectiveness of intercostal cryoneurolysis in patients with pectus excavatum, lateral thoracotomy, post-thoracotomy pain syndrome, traumatic rib fracture and chest wall malignancy. Most studies have demonstrated a reduction in inpatient opioid analgesic use with intercostal nerve cryoablation compared with traditional pain management techniques. In patients requiring lateral thoracotomy, intercostal cryoablation results in decreased opioid analgesic dosage (grade 2A) and improved pain scores (grade 2C) postoperatively (PICO guidelines).

Finding an effective and at the same time simple strategy for pain relief in the early postoperative period in patients undergoing minimally invasive mitral valve surgery is an urgent task; it is advisable to conduct a prospective clinical study with a well-thought-out design in this direction.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent;
* Minimally invasive mitral valve surgery.

Non-inclusion criteria:

* patient refusal;
* pregnancy;
* treatment with antidepressants or epileptic drugs;
* depression, which can significantly affect the perception of pain;
* chronic use of analgesics;
* participation in competing randomized clinical trials.

Exclusion criteria:

- Extended mechanical ventilation, more than 12 hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic consumption | 48 hours after surgery
  Opioid analgesics consumption after surgery, calculated in MME

SECONDARY OUTCOMES:
The intensity of pain | After extubation, 6, 12, 24, 36, 48 hours after surgery
  We will use a visual analogue scale (VAS), that represent the severity of symptoms from 0 "no pain" to 10 "very severe pain".
Dynamics of spirography (FEV1, FVC) | before surgery, 48 hours after surgery, before the patient's discharge
Frequency of side effects (nausea, vomiting, etc.) | 48 hours after surgery
Need for inotropic/vasopressor support | during surgery and in the ICU
  yes/no
Duration of mechanical ventilation | 12 hours
  number of hours
Duration of ICU stay | 10 days
  number of days
Duration of hospital stay | 60 days
  number of days
Identifying side effects of intercostal nerve cryoablation procedure (the occurrence of chronic post-thoracotomy pain syndrome, numbness in the right arm and in the area of surgical access) | 2 and 6 months
  follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin Research Institute of Pathology of Circulation, Novosibirsk, Russia

REFERENCES:
- [Background] Navia JL, Cosgrove DM 3rd. Minimally invasive mitral valve operations. Ann Thorac Surg. 1996 Nov;62(5):1542-4. doi: 10.1016/0003-4975(96)00779-5. PMID 8893611
- [Background] Sherazee EA, Chen SA, Li D, Li D, Frank P, Kiaii B. Pain Management Strategies for Minimally Invasive Cardiothoracic Surgery. Innovations (Phila). 2022 May-Jun;17(3):167-176. doi: 10.1177/15569845221091779. Epub 2022 May 6. No abstract available. PMID 35521910
- [Background] Lau WC, Shannon FL, Bolling SF, Romano MA, Sakwa MP, Trescot A, Shi L, Johnson RL, Starnes VA, Grehan JF. Intercostal Cryo Nerve Block in Minimally Invasive Cardiac Surgery: The Prospective Randomized FROST Trial. Pain Ther. 2021 Dec;10(2):1579-1592. doi: 10.1007/s40122-021-00318-0. Epub 2021 Sep 20. PMID 34545530
- [Background] O'Connor LA, Houseman B, Cook T, Quinn CC. Intercostal cryonerve block versus elastomeric infusion pump for postoperative analgesia following surgical stabilization of traumatic rib fractures. Injury. 2023 Nov;54(11):111053. doi: 10.1016/j.injury.2023.111053. Epub 2023 Sep 18. PMID 37741705
- [Background] Maxwell CM, Weksler B, Houda J, Fernando HC. Intercostal Cryoablation During Video-Assisted Lung Resection Can Decrease Postoperative Opioid Use. Innovations (Phila). 2023 Jul-Aug;18(4):352-356. doi: 10.1177/15569845231185583. Epub 2023 Jul 17. PMID 37461202
- [Background] Nelson KM, Vincent RG, Bourke RS, Smith DE, Blakeley WR, Kaplan RJ, Pollay M. Intraoperative intercostal nerve freezing to prevent postthoracotomy pain. Ann Thorac Surg. 1974 Sep;18(3):280-5. doi: 10.1016/s0003-4975(10)64357-3. No abstract available. PMID 4413968
- [Background] Bucerius J, Metz S, Walther T, Doll N, Falk V, Diegeler A, Autschbach R, Mohr FW. Pain is significantly reduced by cryoablation therapy in patients with lateral minithoracotomy. Ann Thorac Surg. 2000 Sep;70(3):1100-4. doi: 10.1016/s0003-4975(00)01766-5. PMID 11016387
- [Background] Koons B, Suzuki Y, Cevasco M, Bermudez CA, Harmon MT, Dallara L, Ramon CV, Nottingham A, Ganjoo N, Diamond JM, Christie JD, Localio AR, Cantu E. Cryoablation in lung transplantation: Its impact on pain, opioid use, and outcomes. JTCVS Open. 2022 Nov 25;13:444-456. doi: 10.1016/j.xjon.2022.11.005. eCollection 2023 Mar. PMID 37063121
- [Background] Bolotin G, Lazarovici H, Uretzky G, Zlotnick AY, Tamir A, Saute M. The efficacy of intraoperative internal intercostal nerve block during video-assisted thoracic surgery on postoperative pain. Ann Thorac Surg. 2000 Dec;70(6):1872-5. doi: 10.1016/s0003-4975(00)01757-4. PMID 11156086
- [Background] Mamoun NF, Lin P, Zimmerman NM, Mascha EJ, Mick SL, Insler SR, Sessler DI, Duncan AE. Intravenous acetaminophen analgesia after cardiac surgery: A randomized, blinded, controlled superiority trial. J Thorac Cardiovasc Surg. 2016 Sep;152(3):881-889.e1. doi: 10.1016/j.jtcvs.2016.04.078. Epub 2016 May 5. PMID 27236864
- See also: Bogachev-Prokofiev A. V. et al. Pathology of the mitral valve in connective tissue dysplasia — https://doi.org/10.15829/1560-4071-2016-11-81-86
- See also: Hoan D. T. et al. Continuous Unilateral Erector Spinae Plane Block versus Intravenous Analgesia in Minimally Invasive Cardiac Surgery: A Randomized Controlled Trial — https://doi.org/10.3889/oamjms.2022.9071
- See also: Borys M. et al. Erector spinae-plane block as an analgesic alternative in patients undergoing mitral and/or tricuspid valve repair through a right mini-thoracotomy-an observational cohort study — https://doi.org/10.5114/wiitm.2019.85396
- See also: Cha P. I. et al. Efficacy of intercostal cryoneurolysis as an analgesic adjunct for chest wall pain after surgery or trauma: systematic review — https://doi.org/10.1136/tsaco-2021-000690

DOCUMENTS (1):
  • Study Protocol (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT06443931/Prot_001.pdf